CLINICAL TRIAL: NCT01815788
Title: Evaluation of Efficacy and Patient Acceptance of Sound Amplifier Téo First, in Mild and Moderate Presbycusis Patient 60 Years of Age and Older, With no Previous Hearing Aid.
Acronym: TEO FIRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-PP-17
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Mild and Moderate Presbycusis
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Teo first (Experimental): * Mild and moderate presbycusis (20 to 50 dB average hearing loss at 500, 1000, 2000 Hz and 4000 Hz)
  * Patient 60 years of age and older,
  * No previous hearing aid
  Interventions: Device: Use of a personal sound amplifying device = TeoFirst

INTERVENTIONS:
Device: Use of a personal sound amplifying device = TeoFirst

SUMMARY:
A personal sound amplifying device (PASP) like Teo First is a wearable electronic product that is not intended to compensate for impaired hearing, but rather is intended for non-hearing impaired consumers to amplify sounds in the environment for a number of reasons, such as for recreational activities. Nevertheless, a lot of mild and moderate impaired hearing people don't want to buy and wear all day a real hearing aid.

The goal of our study is to evaluate the benefit of such a device for mild and moderate presbycusis patient 60 years of age and older, with no previous hearing aid.

ELIGIBILITY:
Inclusion Criteria:

* Wish to increase hearing
* Moral commitment to use the device
* Ability to understand the study
* Mild and moderate presbycusis (20 to 50 dB average hearing loss at 500, 1000, 2000 Hz and 4000 Hz)
* Patient 60 years of age and older,
* No previous hearing aid

Exclusion Criteria:

* Inability to use the device
* Previous use of a hearing aid
* local intolerance

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Audiometric tests (pure tone and speech) in silence and noise, with and without Teofirst | 7 to 15 days after the first use of Teofirst

SECONDARY OUTCOMES:
audiometric and mental tests | D7 to 15 and D 40
  * Glasgow Hearing Aid Benefit Profile (GHABP)
  * Acceptability and use questionnaire
  * ANL (Acceptable Noise Level) test
  * Mini Mental State Examination
  * Instrumental Activities of Daily Living (IADL)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GUEVARA, PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

REFERENCES:
- [Derived] Sacco G, Gonfrier S, Teboul B, Gahide I, Prate F, Demory-Zory M, Turpin JM, Vuagnoux C, Genovese P, Schneider S, Guerin O, Guevara N. Clinical evaluation of an over-the-counter hearing aid (TEO First(R)) in elderly patients suffering of mild to moderate hearing loss. BMC Geriatr. 2016 Jul 9;16:136. doi: 10.1186/s12877-016-0304-4. PMID 27392722